CLINICAL TRIAL: NCT07140588
Title: Pilot Study of Intraoperative Somatic-Autonomic Nerve Grafting Technique to Preserve Erectile Function in Patients With Bladder Cancer Undergoing Radical Cystectomy
Brief Title: Pilot Study of a New Nerve Grafting Method During Bladder Cancer Surgery to Help Preserve Erections.
Acronym: NR-RC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Victor McPherson, Assistant Professor Division of Urology, Department of Surgery McGill University, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2026-4614
Record Dates: First submitted 2025-07-25; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Bladder Cancer Requiring Cystectomy; Erectile Dysfunction Following Radical Prostatectomy
Keywords: Bladder cancer; Nerve grafting; The genitofemoral nerve; radical cystectomy; radical prostatectomy; Erectile function; International Index of Erectile Function-5; Short Form McGill Pain Questionnaire; Clinical Evolution of Erectile Function
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nerve Restoring Radical Cystectomy. (Experimental): Patients undergoing radical cystectomy will receive a novel NR-RC procedure using a genitofemoral nerve graft to enhance erectile function recovery.
  Interventions: Procedure: Patients undergoing radical cystectomy will receive a novel NR-RC procedure using a genitofemoral nerve graft to enhance erectile function recovery.

INTERVENTIONS:
Procedure: Patients undergoing radical cystectomy will receive a novel NR-RC procedure using a genitofemoral nerve graft to enhance erectile function recovery. — Patients undergoing radical cystectomy will receive a novel NR-RC procedure using a genitofemoral nerve graft to enhance erectile function recovery.

SUMMARY:
This pilot study will evaluate the safety and 1-year erectile function recovery in 10 patients undergoing a novel Nerve Restoring Radical Cystectomy (NR-RC), which includes a genitofemoral nerve graft. Erectile function will be assessed using IIEF-5, SF-MPQ, and CEEF questionnaires at baseline and at multiple post-operative intervals (4 weeks, 3, 6, 12, and 18 months). Safety will be monitored through peri- and post-operative complications, and additional demographic and clinical data will be collected for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing standard of care radical cystectomy for bladder cancer
* Patients must have preoperative erectile function with a baseline IIEF score of ≥17

Exclusion Criteria:

* Patients with previous pelvic surgery
* Patients with previous pelvic radiotherapy
* Patients aged < 18 years at diagnosis
* Legally incapable patients
* Patients who are unable to complete questionnaires and have no companion to help complete them
* Patients undergoing a concomitant cancer surgery
* Patients with pre-existing neurologic disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Adverse events measured by the Clavian-Dindo classification | Through study completion, an average of 18 months (5 different time points)
  The primary outcome is specifically the safety of the operation measured by adverse events as defined by the Clavian-Dindo classification. The measurement varies from Grade I (Best possible outcome) to Grade V (Worst possible outcome). Grade I Deviation from normal p/o course. No pharmacological or surgical treatment, endoscopic or radiological interventions were required. Acceptable therapeutic drugs such as anti-emetics, antipyretics, analgesics, diuretics,electrolytes, physiotherapy. Wound infections, small abscess requiring incision at bedside. Grade II Normal course altered. Pharmacological management other than in Grade I. Blood transfusions and total parenteral nutrition are also included. Grade III Complications that require intervention of various degrees. Grade IV Complications threatening life of patients (including Central Nervous System complications), requiring Intensive Treatment Unit support. Grade V Death of a patient

SECONDARY OUTCOMES:
Clinical Evolution of Erectile Function (CEEF) | 4 weeks post- NR-RC
  A one question visual questionnaire evaluating the erectile function, from 0 (no erection - Worst Possible Outcome) to 10 (sexual intercourse - Best Possible Outcome).
Clinical Evolution of Erectile Function (CEEF) | 3 months post- NR-RC
  A one question visual questionnaire evaluating the erectile function, from 0 (no erection - Worst Possible Outcome) to 10 (sexual intercourse - Best Possible Outcome).
Clinical Evolution of Erectile Function (CEEF) | 6 months post- NR-RC
  A one question visual questionnaire evaluating the erectile function, from 0 (no erection - Worst Possible Outcome) to 10 (sexual intercourse - Best Possible Outcome).
Clinical Evolution of Erectile Function (CEEF) | 12 months post- NR-RC
  A one question visual questionnaire evaluating the erectile function, from 0 (no erection - Worst Possible Outcome) to 10 (sexual intercourse - Best Possible Outcome).
Clinical Evolution of Erectile Function (CEEF) | 18 months post- NR-RC
  A one question visual questionnaire evaluating the erectile function, from 0 (no erection - Worst Possible Outcome) to 10 (sexual intercourse - Best Possible Outcome).
International Index of Erectile Function-5 (IIEF-5) | 4 weeks post- NR-RC
  The IIEF-5 is used to determine the prevalence of erectile dysfunction (ED) in a non-selected population using the abridged 5-item version of the International Index of Erectile Function (IIEF-5) as a diagnostic tool. Each answer has a score from 1 (very low) to 5 (very high). The sum of all the answers gives a final result of 1-7 (Severe ED - Worst Outcome), 8-11 (Moderate ED), 12-16 (Mild-moderate ED), 17-21 (Mild ED) and 22-25 (No ED - Best Outcome).
International Index of Erectile Function-5 (IIEF-5) | 3 months post- NR-RC
  The IIEF-5 is used to determine the prevalence of erectile dysfunction (ED) in a non-selected population using the abridged 5-item version of the International Index of Erectile Function (IIEF-5) as a diagnostic tool. Each answer has a score from 1 (very low) to 5 (very high). The sum of all the answers gives a final result of 1-7 (Severe ED - Worst Outcome), 8-11 (Moderate ED), 12-16 (Mild-moderate ED), 17-21 (Mild ED) and 22-25 (No ED - Best Outcome).
International Index of Erectile Function-5 (IIEF-5) | 6 months post- NR-RC
  The IIEF-5 is used to determine the prevalence of erectile dysfunction (ED) in a non-selected population using the abridged 5-item version of the International Index of Erectile Function (IIEF-5) as a diagnostic tool. Each answer has a score from 1 (very low) to 5 (very high). The sum of all the answers gives a final result of 1-7 (Severe ED - Worst Outcome), 8-11 (Moderate ED), 12-16 (Mild-moderate ED), 17-21 (Mild ED) and 22-25 (No ED - Best Outcome).
International Index of Erectile Function-5 (IIEF-5) | 12 months post- NR-RC
  The IIEF-5 is used to determine the prevalence of erectile dysfunction (ED) in a non-selected population using the abridged 5-item version of the International Index of Erectile Function (IIEF-5) as a diagnostic tool. Each answer has a score from 1 (very low) to 5 (very high). The sum of all the answers gives a final result of 1-7 (Severe ED - Worst Outcome), 8-11 (Moderate ED), 12-16 (Mild-moderate ED), 17-21 (Mild ED) and 22-25 (No ED - Best Outcome).
International Index of Erectile Function-5 (IIEF-5) | 18 months post- NR-RC
  The IIEF-5 is used to determine the prevalence of erectile dysfunction (ED) in a non-selected population using the abridged 5-item version of the International Index of Erectile Function (IIEF-5) as a diagnostic tool. Each answer has a score from 1 (very low) to 5 (very high). The sum of all the answers gives a final result of 1-7 (Severe ED - Worst Outcome), 8-11 (Moderate ED), 12-16 (Mild-moderate ED), 17-21 (Mild ED) and 22-25 (No ED - Best Outcome).
Short Form McGill Pain Questionnaire (SF-MPQ) | 4 weeks post- NR-RC
  The SF-MPQ was designed to measure post-surgical pain. The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe. Three pain scores are derived from the sum of the intensity rank values of the words chosen for sensory, affective and total descriptors. The sum of the scores gives a range of outcomes; a score of 0 (no pain - Best Possible Outcome) to a score of 45 (Most severe pain - Worst Possible Outcome)
Short Form McGill Pain Questionnaire (SF-MPQ) | 3 months post- NR-RC
  The SF-MPQ was designed to measure post-surgical pain. The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe. Three pain scores are derived from the sum of the intensity rank values of the words chosen for sensory, affective and total descriptors. The sum of the scores gives a range of outcomes; a score of 0 (no pain - Best Possible Outcome) to a score of 45 (Most severe pain - Worst Possible Outcome)
Short Form McGill Pain Questionnaire (SF-MPQ) | 6 months post- NR-RC
  The SF-MPQ was designed to measure post-surgical pain. The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe. Three pain scores are derived from the sum of the intensity rank values of the words chosen for sensory, affective and total descriptors. The sum of the scores gives a range of outcomes; a score of 0 (no pain - Best Possible Outcome) to a score of 45 (Most severe pain - Worst Possible Outcome)
Short Form McGill Pain Questionnaire (SF-MPQ) | 12 months post- NR-RC
  The SF-MPQ was designed to measure post-surgical pain. The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe. Three pain scores are derived from the sum of the intensity rank values of the words chosen for sensory, affective and total descriptors. The sum of the scores gives a range of outcomes; a score of 0 (no pain - Best Possible Outcome) to a score of 45 (Most severe pain - Worst Possible Outcome)
Short Form McGill Pain Questionnaire (SF-MPQ) | 18 months post- NR-RC
  The SF-MPQ was designed to measure post-surgical pain. The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe. Three pain scores are derived from the sum of the intensity rank values of the words chosen for sensory, affective and total descriptors. The sum of the scores gives a range of outcomes; a score of 0 (no pain - Best Possible Outcome) to a score of 45 (Most severe pain - Worst Possible Outcome)